CLINICAL TRIAL: NCT03594604
Title: Norethindrone Versus Combined Oral Contraceptive Pills for the Delay of Menstruation
Brief Title: Norethindrone for the Delay of Menstruation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Maurice-Andre Recanati, Assistant Professor, Clinical Educator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 040818M1
Record Dates: First submitted 2018-06-18; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Menstrual Flow Altered
Keywords: norethindrone
MeSH Terms: interventions — Norethindrone; Norethindrone Acetate; Contraceptives, Oral; Contraceptives, Oral, Combined

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive oral contraceptive pills or norethindrone
Who Masked: Investigator
Masking Description: Patients will be randomized to receive oral contraceptive pills or norethindrone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norethindrone (Experimental): Delaying menstruation using Norethindrone 5mg three times daily in women who desire postponement of their period for social or personal reasons.
  Interventions: Drug: Norethindrone
- Oral Contraceptive Pills (Active Comparator): Women who desire postponing their periods are typically treated with oral contraceptive pills, the current standard of care.
  Interventions: Drug: oral contraceptive pill

INTERVENTIONS:
Drug: Norethindrone — Women desiring to postpone their periods may be randomized to norethindrone 5mg three times daily.
  Other Names: (Aygestin)
  Arms: Norethindrone
Drug: oral contraceptive pill — Women desiring to postpone their periods may be randomized to daily oral contraceptive pills.
  Other Names: Combined oral contraceptive pill
  Arms: Oral Contraceptive Pills

SUMMARY:
Comparison of oral contraceptive pills versus norethindrone to delay menstuation.

DETAILED DESCRIPTION:
Many women ask the OBGYN for help in delaying a poorly timed period in order to participate in events that menstruation would normally interfere with. While most OBGYNs prescribe combined oral contraceptives for this purpose, this method often results in unpredictable spotting, especially at the beginning of therapy. Norethindrone, a progesterone agonist, inhibits ovulation through its antagonistic effect at the anterior pituitary, preventing the release of LH. Additionally, it thickens cervical mucus to inhibit sperm migration into the uterine cavity . Norethindrone downregulates estrogen receptors on the endometrium lining preventing endometrial proliferation, enhancing glandular secretion, and maintaining endometrium integrity. Therefore, norethindrone is well suited in preventing the endometrium from breakdown and preventing menstrual bleeding. Indeed, many OBGYNs have consistently used it for this purpose in women who desire to remain fertile. The intention of our study was to compare norethindrone to birth control pills in order to determine the effectiveness at suppressing bleeding and spotting, compare side effect profiles and to find a method allowing women to freely and comfortably participate in their life events.

OBJECTIVES:

1. Determine if norethindrone can delay menstruation without breakthrough bleeding
2. Compare norethindrone with oral contraceptive pills for delaying menstruation
3. Compare patient satisfaction of each method
4. Compare side effect profiles of each method

ELIGIBILITY:
Inclusion Criteria:

* female, age 18-45, regular periods, desires to postpone menstrual period,

Exclusion Criteria:

* fibroids, irregular menstrual cycle, endometrial polyps, BMI>30

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females menstruate
Enrollment: 17 (Actual)
Dates: Start 2007-06-15 (Actual); Primary Completion 2007-12-15 (Actual); Study Completion 2007-12-15 (Actual)

PRIMARY OUTCOMES:
breakthrough bleeding on treatment | at 2 weeks from starting therapy
  comparison of breakthrough bleeding between oral contraceptives and norethindrone

SECONDARY OUTCOMES:
Likelihood of recommending this method or using it again | at 2 weeks from starting therapty
  A questionnaire given to the patient at 2 weeks from starting therapy and containing the question "on a scale from 1-5 (5 most likely) how likely are you to recommend this method to a friend or using it again yourself".
Adverse effects | at 2 weeks from starting therapy
  measurement of side effects from norethindrone therapy

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Recanati, Principal Investigator — St. Vincents Catholic Medical Centers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attia AM, Ibrahim MM, Abou-Setta AM. Role of the levonorgestrel intrauterine system in effective contraception. Patient Prefer Adherence. 2013 Aug 9;7:777-85. doi: 10.2147/PPA.S36948. eCollection 2013. PMID 23990713
- [Result] Yairi-Oron Y, Rabinson J, Orvieto R. A simplified approach to religious infertility. Fertil Steril. 2006 Dec;86(6):1771-2. doi: 10.1016/j.fertnstert.2006.05.050. Epub 2006 Oct 30. PMID 17074351
- [Result] Chertok IR, Zimmerman DR, Taragin S, Silverman Z, Hallak M. Implications of endometriosis for women who observe Jewish law (halakha). Isr Med Assoc J. 2005 Feb;7(2):71-4. PMID 15729953
- [Result] Amy JJ, Tripathi V. Contraception for women: an evidence based overview. BMJ. 2009 Aug 7;339:b2895. doi: 10.1136/bmj.b2895. No abstract available. PMID 19666684
- [Derived] Dean J, Kramer KJ, Akbary F, Wade S, Huttemann M, Berman JM, Recanati MA. Norethindrone is superior to combined oral contraceptive pills in short-term delay of menses and onset of breakthrough bleeding: a randomized trial. BMC Womens Health. 2019 May 28;19(1):70. doi: 10.1186/s12905-019-0766-6. PMID 31138184